CLINICAL TRIAL: NCT05111886
Title: Effectiveness of an Online Parenting Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Mehus, C; R34MH124690 (NIH)
Record Dates: First submitted 2021-10-14; First posted 2021-11-08 (Actual); Results first posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Behavior Problem; Behavior, Child; Parents; Parent-Child Relations
Keywords: Parent program, GenerationPMTO; Primary care referral, pediatric referral; Primary care communication skills training; Online delivery; Brief interventions; Parents of 3-5 year old children; Behavior concerns; Parent behavior; Child externalizing, child internalizing; Acceptability, appropriateness, feasibility
MeSH Terms: conditions — Mental Disorders; Child Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Primary Care Personnel Training (Experimental): Primary care personnel within two Federally Qualified Health Center (FQHC) primary care clinics will be randomly assigned to receive communication skills training or a control condition.
  Interventions: Behavioral: Communication Skills Training; Diagnostic Test: Survey of Experience
- Primary Care Personnel Training Control (Active Comparator): Primary care personnel within two Federally Qualified Health Center (FQHC) primary care clinics will be randomly assigned to receive communication skills training or a control condition. Control group personnel will receive a written description of the referral process but no training.
  Interventions: Behavioral: Written Referral Process; Diagnostic Test: Survey of Experience
- Parents eHealth GenPMTO (Experimental): Parents of 3- to 5-year-olds who receive services from primary care personnel at an Federally Qualified Health Center (FQHC) primary care clinic. Primary care personnel will refer parents of child with externalizing or internalizing behaviors to study therapists. Parents may be assigned to GenPMTO or control after referral.
  Interventions: Behavioral: eHealth GenPMTO; Diagnostic Test: Survey of Experience
- Parents Control (Active Comparator): Parents of 3- to 5-year-olds who receive services from primary care personnel at an Federally Qualified Health Center (FQHC) primary care clinic. Primary care personnel will refer parents of child with externalizing or internalizing behaviors to study therapists. Parents may be assigned to GenPMTO or control after referral.
  Interventions: Behavioral: One Session Education about Resources; Diagnostic Test: Survey of Experience
- Therapists (Other): Community therapists trained to deliver GenPMTO.
  Interventions: Diagnostic Test: Survey of Experience

INTERVENTIONS:
Behavioral: Communication Skills Training — The training will focus on communication skills based on key constructs in the Health Belief Model and motivation/resistance research (described in section A3), the training will focus on: (1) conveying the benefits of parenting programs, (2) knowledge of and responses to common perceived barriers to attending parenting programs, and (3) skills and strategies to effectively motivate and refer parents in ways that are least likely to elicit resistance. The in-person training will last 60-90 minutes. It will include a theoretical background and experiential learning; each step of the referral process will be demonstrated and role-played. The investigators will work to ensure that personnel receive continuing education credits for the training.
  Arms: Primary Care Personnel Training
Behavioral: eHealth GenPMTO — The GenPMTO is delivered over the phone (not online). This version is up to 6 sessions in length. This brief eHealth version of GenPMTO will be delivered through community therapists. The program will be delivered one-on-one (i.e., between a therapist and a parent or couple).
  Arms: Parents eHealth GenPMTO
Behavioral: Written Referral Process — A written summary and process map of the referral process, modeled on the Institute for Healthcare Improvement (IHI) 9-step process for "closing the loop" on referrals.
  Arms: Primary Care Personnel Training Control
Behavioral: One Session Education about Resources — One online or phone conversation with the therapist in which the therapist guides the parent to the following resources: (a) a book, Raising Cooperative Kids, by GenPMTO co-developer Marion Forgatch; (b) a website, behaviorchecker.org, which includes behavioral "prescriptions" for common behavior issues; and (c) information about Early Childhood and Family Education classes, which are provided for free in Minnesota through public schools.
  Arms: Parents Control
Diagnostic Test: Survey of Experience — Satisfaction with referral process

SUMMARY:
Child and adolescent behavioral health problems are related to the leading causes of youth morbidity and mortality. Parent-focused preventive interventions, such as GenerationPMTO (GenPMTO), effectively prevent behavioral health problems such as depression and conduct disorders. Unfortunately, parenting programs are not widely available nor well-attended. Pediatric primary care (PC) is a non-stigmatizing setting with nearly universal reach and, therefore, an ideal access point to increase availability. However, PC personnel are not trained to address behavioral health topics. Also, typical referral practices are inadequate. There is a need to develop effective referral practices in conjunction with increasing availability. There are also logistical barriers to attending in-person parenting programs, like the need for childcare and a large time-commitment. There is a need to overcome these logistical barriers with more accessible programs. The long-term goal is to prevent significant behavioral health problems by increasing access to GenPMTO.

DETAILED DESCRIPTION:
Specifically, the investigators propose engaging parents of 3 to 5-year-olds with moderate externalizing or internalizing symptoms through pediatric primary care (PC); PC personnel will refer parents to a community therapist who will deliver a novel brief eHealth (i.e. online video-chat) model of GenPMTO. Collaborating clinics are part of a Federally Qualified Health Center (FQHC), allowing for access to an under-served population of parents.

The primary objective of this project is to test a brief eHealth version of GenPMTO, delivered to parents online by community therapists (Aim 3). Brief online delivery can overcome logistical barriers, thereby increasing access while maintaining effectiveness. An additional objective is to develop (Aim 1) and test (Aim 2) a brief training for PC personnel and a referral process to equip them to effectively refer parents to eHealth GenPMTO, thereby increasing access to needed services through effective engagement in a trusted setting.

To achieve these objectives, the following aims will be completed. Aim 1 is a development phase to inform Aim 2 components. Aims 2 and 3 run concurrently in the study; the order of the aims reflects the patient flow.

Aim 1: Develop a referral process and a training for PC personnel by gathering mixed-method expert and stakeholder input and feedback. The investigators will present a proposed referral process and PC personnel training, and solicit feedback via the Nominal Group Technique from four expert groups: (1) researchers and implementers (n=6) with experience delivering other parenting interventions though primary care in the U.S., (2) primary care personnel (n=9) from FQHC primary care clinics, (3) personnel from British Columbia (n=6) who have implemented brief GenPMTO over the telephone with parents referred by primary care, and (4) parents (n=6) who receive care from an FQHC. One key question that will be addressed is which PC personnel (e.g., provider, nurse) is best suited to have the referring conversation with parents and receive the training.

Aim 2: Evaluate the referral process and conduct a pilot test of the PC personnel training within FQHC clinics. PC personnel (n=35) within two FQHC primary care clinics will be randomly assigned to receive communication skills training or a control condition. Control group personnel will receive a written description of the referral process but no training. Aim 2a: Using a sequential mixed-methods approach with PC personnel, the investigators will evaluate the acceptability and appropriateness of the referral process and the training. The investigators will also interview parents who do not complete a referral (n=10) to examine the acceptability of the referral process and identify remaining barriers to engagement. Aim 2b: The investigators will pilot test the effectiveness of the training to increase PC personnel's communication skills. The investigators will also use EHR data to pilot test the effect of the training on parent engagement in GenPMTO by comparing the rates of referral and engagement among patients who had an appointment with personnel in the training arm to those seeing control personnel.

Aim 3: Pilot test a brief, eHealth version of GenerationPMTO for moderate externalizing or internalizing symptoms. The personnel described in Aim 2 will refer parents to GenPMTO. Aim 3a: With the referred parents, the investigators will conduct a pilot RCT to examine change in parents' (n=60) parenting locus of control, self-reported parenting behaviors, and child externalizing and internalizing, all of which have been shown to predict later changes in child behavioral health outcomes. The investigators will examine the mediating effect of parenting changes on changes in child outcomes. These effect sizes will also be compared to effect sizes from other GenPMTO studies to determine if this preliminary assessment aligns with findings from other versions of GenPMTO. Aim 3b: Using a sequential mixed-methods approach, the investigators will assess the acceptability, feasibility, and appropriateness of brief, eHealth GenPMTO among therapists (n=15) and a sub-sample of parents (n=14).

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible for Aim 1 if they are:

* Able to speak English
* Able to participate in the focus group

Participants are eligible for Aim 2 if they are:

* Primary care personnel who are currently practicing in a collaborating clinic
* Therapists who are eligible for reimbursement from insurance and Medicaid
* Parents who are:

  1. Referred to a therapist by their providers
  2. Have the ability to speak English or Spanish, and
  3. Are a primary caregiver for a child between the ages of 3 and 5 years old

Exclusion Criteria:

* None

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Mehus, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be deposited in NIH data repository.
Supporting Information: SAP
Time Frame: 3 years

REFERENCES:
- [Background] Clerkin SM, Marks DJ, Policaro KL, Halperin JM. Psychometric properties of the Alabama parenting questionnaire-preschool revision. J Clin Child Adolesc Psychol. 2007 Mar;36(1):19-28. doi: 10.1080/15374410709336565. PMID 17206878
- [Background] Forgatch MS, Patterson GR, DeGarmo DS. Evaluating fidelity: predictive validity for a measure of competent adherence to the Oregon model of parent management training. Behav Ther. 2005;36(1):3-13. doi: 10.1016/s0005-7894(05)80049-8. PMID 16718302
- [Background] Helfrich CD, Li YF, Sharp ND, Sales AE. Organizational readiness to change assessment (ORCA): development of an instrument based on the Promoting Action on Research in Health Services (PARIHS) framework. Implement Sci. 2009 Jul 14;4:38. doi: 10.1186/1748-5908-4-38. PMID 19594942
- [Background] Lovejoy MC, Verda MR, Hays CE. Convergent and discriminant validity of measures of parenting efficacy and control. J Clin Child Psychol. 1997 Dec;26(4):366-76. doi: 10.1207/s15374424jccp2604_5. PMID 9418175
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Kamphaus, R. W. & Reynolds, C. R. (2015). BASC 3 Behavioral and Emotional Screening System Manual. Pearson PsychCorp.
- [Background] Mehus, C., Ballard, J., Driscoll, J., Sargeant, L., & Exsted, M. (2025). Support and Guide: Observational Coding Scale Manual for Primary Care Clinician Conversations with Parents. University of Minnesota Digital Conservancy. Retrieved from https://hdl.handle.net/11299/276913

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Primary Care Personnel Training | Primary Care Personnel Training Control | Parents eHealth GenPMTO | Parents Control | Therapists
Started | 21 | 14 | 23 | 20 | 16
Completed | 21 | 14 | 23 | 16 | 16
Not Completed | 0 | 0 | 0 | 4 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Primary Care Personnel Training | Primary Care Personnel Training Control | Parents eHealth GenPMTO | Parents Control | Therapists | Total
Number analyzed (Participants) | 21 | 14 | 23 | 20 | 16 | 94
Age, Categorical [Count of Participants; unit: Participants] — Population: The 'Number analyzed' reported for age reflects the total number who reported their age (e.g., 14 clinicians in the experimental condition of 21 total, 12 clinicians in the control condition of 14 total, 23 parent participants in the eGen condition of 23 total, 20 participants in the control condition of 20 total, and 16 participants in the therapist condition of 16 total.
  Participants
    number analyzed (Participants) | 14 | 12 | 23 | 20 | 16 | 85
    <=18 years | 0 | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 13 | 12 | 23 | 19 | 16 | 83
    >=65 years | 1 | 0 | 0 | 1 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The 'Number analyzed' reported for sex reflects the total number who reported their sex (e.g., 16 clinicians in the experimental condition of 21 total, 12 clinicians in the control condition of 14 total, 23 parent participants in the eGen condition of 23 total, 20 participants in the control condition of 20 total, and 15 participants in the therapist condition of 16 total.
  Participants
    number analyzed (Participants) | 16 | 12 | 23 | 20 | 15 | 86
    Female | 14 | 8 | 22 | 19 | 15 | 78
    Male | 2 | 4 | 1 | 1 | 0 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 0 | 0 | 2
  Asian | 2 | 2 | 0 | 0 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 4 | 4 | 12
  White | 11 | 8 | 10 | 7 | 6 | 42
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 7 | 3 | 9 | 9 | 5 | 33

OUTCOME MEASURES:

1. Primary Outcome: Aim 3: Change in Behavioral Assessment System Child Score
Description: Outcome is reported as the difference in pre- and post-intervention Externalizing Risk Scores, a subscale from the Behavior Assessment System for Children (3rd Edition, Parent Report Form - Preschool), which measures externalizing, internalizing, and adaptive behaviors. The Externalizing Risk Scores subscale measures externalizing behaviors the sum of using 9 items with a four-choice response format, for a raw Externalizing Risk Score range of 0-27. Higher scores indicate worse levels of externalizing behavior functioning. Scores of 0-10 are in the normal risk range, scores of 11-19 are elevated, and scores of 20 or above are extremely elevated. This is administered to parents before and after the intervention window (8 week separation). The change score was calculated as the value at 8 weeks minus value at baseline.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parents eHealth GenPMTO | Parents Control
Number analyzed (Participants) | 23 | 16
score on a scale | -3.17 (7.51) | 0.13 (8.76)

2. Primary Outcome: Aim 3: Change in Alabama Parenting Questionnaire
Description: Outcome is reported as the difference in total scale score on the Alabama Parenting Questionnaire (preschool version) (Clerkin et al., 2007). This questionnaire contains 32 items rated on a 5-point scale ranging from "Never" to "Always." Total scores range from 32 to 160 with higher score indicating more involvement and positive parenting. This is administered to parents before and after the intervention window (8 week separation).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parents eHealth GenPMTO | Parents Control
Number analyzed (Participants) | 23 | 16
score on a scale | -0.65 (1.94) | -0.13 (1.41)

3. Primary Outcome: Aim 3: Change in Parent Locus of Control
Description: Outcome is reported as the difference in total scores on the Parent Locus of Control measure (Lovejoy et al., 1997). This measure contains 24 items rated on a 5-point scale from strongly disagree (1) to strongly agree (5). Scores range from 24 to 120. High scores on the scale indicate an external locus of parenting control and low scores indicate an internal locus. This is administered to parents before and after the intervention window (8 week separation).
Time Frame: 8 weeks
Population: In the active comparator: parents control condition, 1 person was missing data (1/16)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parents eHealth GenPMTO | Parents Control
Number analyzed (Participants) | 23 | 15
score on a scale | 3.78 (8.05) | 2.47 (7.98)

4. Primary Outcome: Aim 2: Percentage of Completed Referrals
Description: Percentage of eligible appointments leading to successful referral.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: % of appts leading to completed referral
Arm/Group | Primary Care Personnel Training | Primary Care Personnel Training Control
Number analyzed (Participants) | 21 | 14
% of appts leading to completed referral | 0.34 (0.94) | 0.15 (0.37)

5. Primary Outcome: Aim 2: Parent Attendance
Description: For each referred caregiver, the number of sessions attended (0-6) was divided by the total possible number of sessions (6), to calculate the percent of sessions attended. The average was then calculated by referring clinician condition (training or control).
Time Frame: 1 year
Population: The percent of sessions attended can only be calculated for clinicians who made at least one referral. Data is analyzed for 12 primary care clinicians in the training condition and 7 primary care clinicians in the control condition. This reflects that 9/21 clinicians in the training condition did not make any referrals, and 7/14 clinicians in the control condition did not make any referrals
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Primary Care Personnel Training | Primary Care Personnel Training Control
Number analyzed (Participants) | 12 | 7
percent | 22.4 (39.0) | 20.0 (36.0)

6. Primary Outcome: Aim 1: Fidelity of Implementation Rating System
Description: Communication skills rating will be measured using the Support and Guide Observational Coding Scale of audio-recorded provider responses to clinical vignettes, a measure adapted from the Fidelity of Implementation Rating System. The scale measures the communication skills of supporting, guiding, confronting (reverse-coded), teaching (reverse-coded), and tone. Each of these components is averaged across the three vignettes on a 0-3 scale (support, guide, confront, teach), or a 0-2 scale (tone). A total scale is then summed for a total scale score range of 0-14, with higher scores indicating greater communication skills. These vignette prompts are administered to providers before and after the pilot year (1 year separation).
Time Frame: 1 year
Population: Audio-recorded responses were missing for 10 of the 21 primary care clinicians in the experimental condition, and 9 of the 14 primary care clinicians in the control condition
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Primary Care Personnel Training | Primary Care Personnel Training Control
Number analyzed (Participants) | 11 | 5
score on a scale | 11.26 (4.53) | 8.9 (2.56)

7. Secondary Outcome: Intervention Acceptability Measure
Description: Average score on the Acceptability of intervention Measure (4 items) (Weiner et al., 2017), which assesses acceptability, or belief that the training is agreeable or satisfactory. Scores are on a 1-5 scale from completely disagree to completely agree, and all four items are averaged for a total score range of 1 to 5. A higher score indicates higher acceptability. This is administered to parents after the intervention window (8 week separation) and to providers and therapists before and after the pilot year (1 year separation).
Time Frame: 8 weeks (Parents) 1 year (Therapists)
Population: Acceptability data was missing for 11 of the 21 primary care clinicians in the experimental condition, and 6 of the 14 primary care clinicians in the control condition. Acceptability data was missing for 5 of the parents in the experimental condition, and 10 of the parents in the control condition. Acceptability data was not missing for any of the therapists.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Primary Care Personnel Training | Primary Care Personnel Training Control | Parents eHealth GenPMTO | Parents Control | Therapists
Number analyzed (Participants) | 10 | 8 | 18 | 6 | 16
score on a scale | 3.3 (0.88) | 3.25 (0.89) | 4.24 (0.8) | 3.13 (1.2) | 4.23 (0.72)

8. Secondary Outcome: Appropriateness Measure
Description: Average score on two appropriateness items assessing appropriateness of time commitment and expected benefit, generated by the researchers. The first item was "My communication with patients will improve as a result of the training," and the second item was "The time commitment for the training was reasonable." Appropriateness refers to perceived fit of the training for the practice setting and patients. Scores are on a 1-5 scale from completely disagree to completely agree. A higher score indicates higher appropriateness. This is administered to providers immediately after the training.
Time Frame: Immediately following training
Population: Appropriateness was only assessed among Primary Care Clinicians in the experimental condition. Of these 21 clinicians, 13 reported on the acceptability.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Primary Care Personnel Training
Number analyzed (Participants) | 13
score on a scale | 4.03 (0.43)

9. Secondary Outcome: Feasibility Measure
Description: Average score on the Feasibility of Intervention Measure (4 items). Feasibility refers to how well the training can be carried out within the agency/clinic setting. Scores are on a 1-5 scale from completely disagree to completely agree. All four items are averaged for a total score range of 1 to 5. A higher score indicates higher feasibility. This is administered to providers and therapists before and after the pilot year (1 year separation).
Time Frame: 1 year
Population: Feasibility was only assessed among Primary Care Clinicians (both arms) and Therapists. Responses to this measure were missing for 11 of the 21 primary care clinicians in the experimental condition, for 6 of the 14 primary care clinicians in the control condition, and for 1 of the 16 therapists. It was not assessed of parents in either arm (active comparator or experimental).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Primary Care Personnel Training | Primary Care Personnel Training Control | Therapists
Number analyzed (Participants) | 10 | 8 | 15
score on a scale | 3.4 (0.74) | 3.44 (0.73) | 4.24 (0.40)

10. Secondary Outcome: Readiness to Change - Patient Preferences Subscale Score
Description: Summed score on the Readiness to Change Assessment, patient preferences (4 items). The patient preferences subscale assesses site readiness to implement new trainings, based on perceived patient preferences. This measure is rated on a 1-5 scale from strongly disagree to strongly agree, with a sixth option for not applicable. Summed scores range from 4 to 20; High scores indicates greater acceptability. This is administered to providers and therapists before and after the pilot year (1 year separation).
Time Frame: 8 weeks, 1 year
Population: Responses to this measure were missing for 10 of the 21 primary care clinicians in the experimental condition, for 2 of the 14 primary care clinicians in the control condition, and for 3 of the 16 therapists. It was not assessed of parents in either arm (active comparator or experimental).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Primary Care Personnel Training | Primary Care Personnel Training Control | Therapists
Number analyzed (Participants) | 11 | 12 | 13
score on a scale | 17.09 (1.58) | 17.25 (1.86) | 16.23 (1.87)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Primary Care Personnel Training | Primary Care Personnel Training Control | Parents eHealth GenPMTO | Parents Control | Therapists
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/14 | 0/23 | 0/20 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/14 | 0/23 | 0/20 | 0/16
Other Adverse Events (participants affected / at risk) | 0/21 | 0/14 | 0/23 | 0/20 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-29): https://cdn.clinicaltrials.gov/large-docs/86/NCT05111886/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-04): https://cdn.clinicaltrials.gov/large-docs/86/NCT05111886/ICF_001.pdf